CLINICAL TRIAL: NCT00335933
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Gabapentin Extended Release (G-ER) Tablets in the Treatment of Patients With Postherpetic Neuralgia
Brief Title: Safety and Efficacy of Gabapentin in Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Depomed (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 81-0045
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2007-08-02 (Estimated); Status verified 2006-06

CONDITIONS: Neuralgia, Postherpetic
Keywords: Postherpetic Neuralgia (PHN)
MeSH Terms: conditions — Neuralgia, Postherpetic

INTERVENTIONS:
Drug: Gabapentin extended-release tablets

SUMMARY:
Gabapentin and pregabalin are treatments for some types of neuropathic pain, including postherpetic neuralgia (PHN). However, these treatments usually need to be taken 3 times a day for effective pain control. The purpose of this study is to determine whether a new gabapentin tablet, which only needs to be taken once or twice a day, is safe and effective for the treatment of postherpetic neuralgia.

DETAILED DESCRIPTION:
The primary study objective is to assess the relative efficacy of G-ER dosed once daily (1800 mg following the evening meal) or twice daily (600 mg AM/1200 mg PM), versus placebo in reducing the mean daily pain score from the baseline week to the end of the efficacy treatment period (Treatment Week 10) in patients with PHN.

Secondary efficacy measures will include changes from baseline in mean weekly sleep interference scores, Short-Form McGill Pain Questionnaire (SF-MPQ), the Neuropathic Pain Scale (NPS), Brief Pain Inventory (BPI), Patient Global Impression of Change (PGIC), and Investigator-Rated Clinical Global Impression of Change (CGIC).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 years or older who have experienced pain for at least 3 months after the healing of a herpes zoster skin rash (typically about 4 months after the rash first appears).
2. Patient has pain intensity score of at least 4 on the 11-point Likert numerical rating scale at screening. Potential patients should not be informed of the pain intensity eligibility criterion prior to screening or randomization.
3. Patients of childbearing potential must have a negative urine pregnancy test at screening/randomization, and must use medically acceptable methods of birth control. Acceptable methods of birth control include oral or transdermal contraceptives, condom, spermicidal foam, intrauterine device (IUD), progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or postmenopausal for ≥ 1 year, must be specified in the patient's case report form (CRF).
4. Patient has a mean baseline week pain intensity score of at least 4 on the 11-point Likert scale at the end of a 1-week pre-treatment period and has completed at least 4 days of daily pain diary entries during the baseline week.
5. Patient must have a minimum washout period of greater than 5 times the half-life of the drug of any of the following medications: benzodiazepines, skeletal muscle relaxants, orally administered steroids, capsaicin, mexiletene, centrally acting analgesics (dextromethorphan, tramadol), opiates, topical lidocaine, anticonvulsants and serotonin and norepinephrine reuptake inhibitors (SNRIs). Anticonvulsants, SNRIs, opiates and benzodiazepines should be tapered appropriately, using product label instructions as a guide.
6. Patients currently treated with gabapentin or pregabalin at screening may be eligible for the study, but must have a tapering period wherein the dose of gabapentin or pregabalin is reduced gradually over a period of at least 7 days plus a 2-day or 3-day washout of gabapentin or pregabalin, respectively, prior to start of the baseline week.

Exclusion Criteria:

1. Patients who have previously not responded to treatment for PHN with gabapentin at doses of ≥ 1200 mg/day or pregabalin at doses ≥ 300 mg/day.
2. Patients who previously experienced dose-limiting adverse effects that prevented titration of gabapentin to an effective dose.
3. Patient is a nursing mother.
4. Patient has hypersensitivity to gabapentin.
5. Patient has had neurolytic or neurosurgical treatment for PHN.
6. Patient has severe pain from causes other than PHN.
7. Patient has used injected anesthetics or steroids within 30 days of baseline.
8. Patient has skin conditions in the area affected by the neuropathy that could alter sensation.
9. Patient is in an immunocompromised state.
10. Patient has an estimated creatinine clearance of < 60 ml/min calculated using the Cockroft Gault method. If the patient fails this criterion, the Investigator may decide to conduct a 24-hour creatinine clearance test. The patient would be allowed to enroll in the study if the 24-hour test result is < 60 ml/min.
11. Patient has had a malignancy within the past 2 years other than basal cell carcinoma.
12. Patient has had gastric reduction surgery.
13. Patient has severe chronic diarrhea, chronic constipation [unless attributed to drugs that will be washed out], uncontrolled irritable bowel syndrome (IBS) or unexplained weight loss.
14. Patient has any abnormal chemistry or hematology results that are deemed by the Investigator to be clinically significant.
15. Patient has a history of substance abuse within the past year.
16. Patient has a history of seizure (except for infantile febrile seizure) or is at risk of seizure due to head trauma.
17. Patient has a history of chronic hepatitis B or C, hepatitis within the past 3 months, or HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2006-05; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary study objective is to assess the relative efficacy of G-ER versus placebo in reducing the average daily pain score from the baseline week to the final week of the efficacy treatment period (Treatment Week 10) in patients with PHN
Daily pain scores will be measured using an electronic diary.

SECONDARY OUTCOMES:
Secondary objectives include assessment of changes from baseline in average daily sleep interference scores.

CONTACTS AND LOCATIONS:
Overall Officials: Bret Berner, Ph.D., Study Director — Sponsor/Depomed, Inc.
Locations (1):
- PPD Development, Austin, Texas, United States

REFERENCES:
- [Derived] Mehta N, Bucior I, Bujanover S, Shah R, Gulati A. Relationship between pain relief, reduction in pain-associated sleep interference, and overall impression of improvement in patients with postherpetic neuralgia treated with extended-release gabapentin. Health Qual Life Outcomes. 2016 Apr 1;14:54. doi: 10.1186/s12955-016-0456-0. PMID 27037091
- [Derived] Wallace MS, Irving G, Cowles VE. Gabapentin extended-release tablets for the treatment of patients with postherpetic neuralgia: a randomized, double-blind, placebo-controlled, multicentre study. Clin Drug Investig. 2010;30(11):765-76. doi: 10.2165/11539520-000000000-00000. PMID 20818838